CLINICAL TRIAL: NCT04260672
Title: Child-Centred Health Dialogue for Primary Prevention of Obesity in Child Health Services
Brief Title: Child-Centred Health Dialogue in Child Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other); Forte (Industry)
Responsible Party: Principal Investigator, Mariette Derwig, Doctoral student, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016721LUC3
Record Dates: First submitted 2020-01-29; First posted 2020-02-07 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Child, Only; Child Obesity; Parents
Keywords: Child nutrition; Child physical activity; Child sleeping routines; Child toothbrushing; Parental feeding practices; Parental self-efficacy
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: A clustered non-blinded randomised controlled trial (RCT) with two arms to determine the effectiveness (including costs and cost effectiveness) of 1) usual care (n = 3015 children) and 2) CCHD (n = 3032 children). The RCT includes 35 Child Health Centres (CHCs), located both in the country side as well as in 2 of the major cities, including areas with diverse social-economic settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child-Centred Health Dialogue (CCHD) (Experimental): The intervention CCHD consists of two parts 1) a universal Child Centred Health Dialog by the CHS-nurse directed in the first place to all 4-year-olds and their families (10 minutes) and 2) a targeted Family Guidance by the CHS-nurse to families where a child is identified with overweight at the age of 4 (60 minutes). All children invites to their regular 5-yrs health visit.
  Interventions: Behavioral: Child Centred Health Dialog (CCHD)
- usual care (No Intervention): Usual care for preschool children identified with overweight and obesity Usual care is performed according to national guidelines that invites all 4-year-olds to a '4-years health visit' including a health conversation. A survey on usual care in the case of identified overweight initial to this study among almost all nurses working at the participating CHCs showed that two thirds of questioned CHS-nurses used to invite families in which the child is identified with overweight for 1 or 2 extra visits outside the usual program. The majority o referred children to a dietician, or to another caregiver. All children invites to their regular 5-yrs health visit.

INTERVENTIONS:
Behavioral: Child Centred Health Dialog (CCHD) — The universal part of CCHD means a structured dialogue between the nurse and the child in presence of its parents using eight illustrations based on the most important practices associated with overweight in preschool children: fruit and vegetables consumption, intake of sweetened beverages and portion size, physical activity, sedentary behaviour tooth brushing and sleep routines. The health dialog is completed by demonstrating the BMI-growth chart to show BMI development to give parents an accurate weight perception, identify overweight and support parental readiness towards a healthy lifestyle.
  When the child is identified with an overweight or obesity, the entire family is invited to participate in the targeted part of CCHD: the Family Guidance, a family consultation based on the evidence based Standardized Obesity Family Therapy (Nowicka, 2011).
  Arms: Child-Centred Health Dialogue (CCHD)

SUMMARY:
Aims: The principal aim of this study is to evaluate a model of Child Centred Health Dialog (CCHD) in Child Health Services (CHS) aiming to promote a healthy lifestyle in families and prevent overweight and obesity in preschool children. The specific aims are to compare CCHD with usual care and to evaluate the effectiveness and cost-effectiveness of the CCHD for all children and specifically for children with overweight at the age of 4 years and to compare parents self-efficacy and feeding practices in families that received either CCHD or usual care Methods: A clustered non-blinded Randomised Control Trial was set up comparing usual care with a structured multicomponent child-centred health dialogue consisting of two parts: 1) a universal part directed to all children and 2) a targeted part for families where the child is identified with overweight.

DETAILED DESCRIPTION:
Obesity in childhood challenges our global health as it affects children's immediate health, educational achievements and quality of life. Research shows that obesity has its roots in the preschool years and that children with obesity are very likely to remain obese as adults and are at risk of developing adult morbidity. Therefore, primary prevention and lifestyle interventions are important in order to promote healthy lifestyle and reduce the likelihood of later obesity. The evidence is strong that the first years of life are critical in establishing good nutrition and physical activity behaviours.

The principal aim of the study is to evaluate a model of Child Centred Health Dialog (CCHD) in Child Health Services (CHS) aiming to promote a healthy lifestyle in families and prevent overweight and obesity in preschool children. Specific aims are to compare CCHD with usual care and to evaluate the effectiveness of the CCHD for all children and specifically for children with overweight at the age of 4 years and to compare parents self-efficacy and feeding practices in families that received either CCHD or usual care and to analyse the cost and cost effectiveness of CCHD, compared to usual care

The study is guided by the Medical Research Councils framework for complex interventions consisting of four key elements: development, feasibility/piloting, evaluation and implementation. In the feasibility phase CCHD proved to be feasible and fewer normal-weight 4-year-olds in the intervention group had developed overweight at the age of 5 compared to the control group and none had developed obesity one year after the intervention. Qualitative interview studies showed that nurses felt more comfortable using the illustrations in the conversation about healthy food habits. The nurses described the children more talkative and more involved when the illustrations were used. Parents felt that they received support, confirmation and guidance on various issues in the health dialogue. Four-year-old children liked to participate actively in CCHD, expressed their views based on their daily life but needed to understand the meaning of the information with which they interacted.

The Swedish Child Health Services (CHS) are free of charge and attended by nearly all families with young children, irrespective of social position or ethnicity. CHS provide a package of health care universally to all children aged 0-5 years and extra health visits are offered according to need. Overweight is a condition, par excellence, that exemplifies the need for this approach. However, evidence-based models that can be used in CHS for the prevention of overweight and the prevention of obesity in case of identified overweight are lacking.

The intervention CCHD was developed based on the following theories: the child's perspective, which puts the child as part of a family in the centre of thinking and practice and health literacy, meaning how people access, understand and use health information in ways which promote and maintain good health.

ELIGIBILITY:
Inclusion Criteria:

* Both intervention and control CHC units will offer all 4-year-old children and their caregivers their regular '4 year health visit'. Nurses working at the intervention CHCs offer families CCHD and nurses working at the Control CHCs offer usual care

Exclusion Criteria:

-

Ages: 42 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6047 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in BMI standard deviation (SD) scores | 12 months post-intervention
  BMI standard deviation (SD) scores also called BMI- z-scores measures relative weight adjusted for child age and sex.

SECONDARY OUTCOMES:
Children's dietary intake, physical activity, sleeping and tooth brushing routines | baseline at four years old, 4 years and 6 months (6 months post-intervention) and 5 years old (12 months post-intervention)
  Both parents fill out a questionnaire at baseline, 6 month and 12 month after the intervention based on the 2013 public health survey of children and parents in Skåne (Köhler 2017) about intake of fruit and vegetables, sweetened beverages, meal (breakfast) habits, number of family mealtimes, number of portions, hours of sedentary behaviors and physical activity, sleeping and tooth brushing routines
Parents self-efficacy for promoting healthy physical activity and dietary behaviors (PSEPAD) in children | baseline at four years old, 4 years and 6 months (6 months post-intervention) and 5 years old (12 months post-intervention)
  The PSEPAD (Bohman, 2013) was developed for use in the context of childhood obesity prevention. The PSEPAD is a self-report measure composed of 12 items, covering three domains of interest in childhood obesity prevention: Parental Self-Efficacy (PSE) for promoting healthy dietary behaviours in children, PSE for promoting healthy physical activity behaviours in children and PSE for limit-setting of unhealthy dietary and physical activity behaviours in children. Caregivers rated the strength of their efficacy beliefs in influencing their preschool children on an 11-point Likert-type scale ranging from 0 to 10, with the following anchors: 0 = not at all, 2 = to a very low degree, 4 = to some degree, 6 = to quite a degree, 8 = to a high degree, 10 = to a very high degree. A total score is achieved by summing up the scores on the 14 items, with a high total score indicating high PSE.
Parental feeding practices concerning parents of preschool-aged children (CFQ) | baseline at four years old, 4 years and 6 months (6 months post-intervention) and 5 years old (12 months post-intervention)
  The Child Feeding Questionnaire (CFQ) measures parental feeding practices and attitudes (Birch 2001). The CFQ contains originally 31 items and measures the following seven factors: Perceived Responsibility (three items), Parent Perceived Weight (four items), Perceived Child Weight (six items), Parents Concern about Child Weight (three items), Parents' feeding practices: Restriction (eight items), Pressure to Eat (four items), and Monitoring (three items). The responses to all items are coded on a 5-point Likert scale ranging from one to five. Validated for Sweden by Nowicka (2014)
Number of referrals for overweight to other caregivers | at 4 years old
  To test the hypothesis that CCHD is less expensive than usual care incremental cost-effectiveness ratios of CCHD compared to usual care will be calculated. The economic analyses will be performed in both a narrow health-care perspective (only health-care costs count) and in a wider societal one (including also effects outside the health-care sector, specifically parents' time costs and loss of production). In both perspectives, three types of effects are used as effectiveness indicators (a) change in BMI, (b) number of extra visits between the regular visits at 4 and 5 years of age and (c) number of referrals for overweight or obesity to other care givers (for example to dietician, General Practitioner, child specialist).
Number of extra visits between the regular visits at 4 and 5 years of age | 12 months post-intervention
  To test the hypothesis that CCHD is less expensive than usual care incremental cost-effectiveness ratios of CCHD compared to usual care will be calculated. The economic analyses will be performed in both a narrow health-care perspective (only health-care costs count) and in a wider societal one (including also effects outside the health-care sector, specifically parents' time costs and loss of production). In both perspectives, three types of effects are used as effectiveness indicators (a) change in BMI, (b) number of extra visits between the regular visits at 4 and 5 years of age and (c) number of referrals for overweight or obesity to other care givers (for example to dietician, General Practitioner, child specialist).
BMI standard deviation (SD) scores 12 months after intervention | 12 months post-intervention
  BMI standard deviation (SD) scores also called BMI- z-scores measures relative weight adjusted for child age and sex.
BMI 12 months after intervention | 12 months post-intervention
  BMI measures relative weight adjusted for child age and sex.
BMI Change | 12 months post-intervention
  BMI measures relative weight adjusted for child age and sex.
Costs | 12 months post-intervention
  health costs and effects outside the health-care sector: parental loss of productivity and costs of transportation, cost for training in intervention

CONTACTS AND LOCATIONS:
Overall Officials: Inger Hallström, Study Chair — Lunds University
Locations (35):
- Sweden (35):
  - Barnavårdscentralen Anderslöv, Anderslöv
  - Barnavårdscentralen Bokskogen, Bara
  - Barnavårdscentralen Kärråkra, Eslöv
  - BVC Brahehälsan Eslöv, Eslöv
  - Adolfsbergs BVC, Helsingborg
  - Barnavårdscentralen Brunnen, Helsingborg
  - BVC Capio Citykliniken Mariastaden, Helsingborg
  - BVC Capio Citykliniken Olympiakliniken, Helsingborg
  - BVC Väla, Helsingborg
  - Familjecentral Fröhuset, Helsingborg
  - Helsingborgs Barnavårdscentral, Helsingborg
  - Barnavårdscentralen Kävlinge, Kävlinge
  - BVC Capio Citykliniken Landskrona, Landskrona
  - BVC Familjecentralen Tellus, Landskrona
  - Barnavårdscentralen Laröd, Laröd
  - Barnavårdscentralen Bunkeflo, Malmo
  - Barnavårdscentralen Granbacksvägen, Malmo
  - Barnavårdscentralen Grankotten, Malmo
  - Barnavårdscentralen Kirseberg, Malmo
  - Barnavårdscentralen Limhamn, Malmo
  - Barnavårdscentralen Lunden, Malmo
  - Barnavårdscentralen Nalle, Malmo
  - Barnavårdscentralen Oxie, Malmo
  - Barnavårdscentralen Sorgenfrimottagningen, Malmo
  - BVC Capio Citykliniken Limhamn, Malmo
  - BVC Capio Citykliniken Singelgatan, Malmo
  - BVC Capio Citykliniken Västra Hamnen, Malmo
  - BVC Familjecentralen Sesam, Malmo
  - BVC Victoria Vård och Hälsa, Malmo
  - Emma Barnavård på Cura, Malmo
  - Familjens Hus Södervärn, Malmo
  - Örestadsklinikens Barnavårdscentral, Malmo
  - Barnavårdscentralen Skurup, Skurup
  - Barnavårdscentralen Familjecentralen Paletten, Staffanstorp
  - BVC Valens Läkargrupp, Trelleborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birch LL, Fisher JO, Grimm-Thomas K, Markey CN, Sawyer R, Johnson SL. Confirmatory factor analysis of the Child Feeding Questionnaire: a measure of parental attitudes, beliefs and practices about child feeding and obesity proneness. Appetite. 2001 Jun;36(3):201-10. doi: 10.1006/appe.2001.0398. PMID 11358344
- [Background] Derwig M, Tiberg I, Bjork J, Hallstrom I. Child-Centred Health Dialogue for primary prevention of obesity in Child Health Services - a feasibility study. Scand J Public Health. 2021 Jun;49(4):384-392. doi: 10.1177/1403494819891025. Epub 2019 Dec 19. PMID 31854251
- [Background] Nowicka P, Sorjonen K, Pietrobelli A, Flodmark CE, Faith MS. Parental feeding practices and associations with child weight status. Swedish validation of the Child Feeding Questionnaire finds parents of 4-year-olds less restrictive. Appetite. 2014 Oct;81:232-41. doi: 10.1016/j.appet.2014.06.027. Epub 2014 Jun 24. PMID 24972134
- [Background] Kohler M, Emmelin M, Rosvall M. Parental health and psychosomatic symptoms in preschool children: A cross-sectional study in Scania, Sweden. Scand J Public Health. 2017 Dec;45(8):846-853. doi: 10.1177/1403494817705561. Epub 2017 Jun 27. PMID 28653567
- [Background] Coyne I, Hallstrom I, Soderback M. Reframing the focus from a family-centred to a child-centred care approach for children's healthcare. J Child Health Care. 2016 Dec;20(4):494-502. doi: 10.1177/1367493516642744. Epub 2016 Jul 25. PMID 27141084
- [Background] Waters E, de Silva-Sanigorski A, Hall BJ, Brown T, Campbell KJ, Gao Y, Armstrong R, Prosser L, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD001871. doi: 10.1002/14651858.CD001871.pub3. PMID 22161367
- [Background] Nowicka P, Flodmark CE. Family therapy as a model for treating childhood obesity: useful tools for clinicians. Clin Child Psychol Psychiatry. 2011 Jan;16(1):129-45. doi: 10.1177/1359104509355020. Epub 2010 Jul 22. PMID 20650975
- [Background] Bohman B, Ghaderi A, Rasmussen F. Psychometric Properties of a New Measure of Parental Self-Efficacy for Promoting Healthy Physical Activity and Dietary Behaviors in Children. European Journal of Psychological Assessment. 2013:291.
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Hakansson L, Derwig M, Olander E. Parents' experiences of a health dialogue in the child health services: a qualitative study. BMC Health Serv Res. 2019 Oct 30;19(1):774. doi: 10.1186/s12913-019-4550-y. PMID 31666057
- See also: illustrations used in the universal part of CCHD — https://www.rikshandboken-bhv.se/metoder--riktlinjer/halsosamtal-om-levnadsvanor/grunda-sunda-vanor---pedagogiskt-bildmaterial/